CLINICAL TRIAL: NCT03825692
Title: A Multi-center, Randomized, Double-Blind, Placebo-Controlled Parallel Group Clinical Trial of Zhizhu Kuanzhong Capsule in Treating Patients With Postprandial Distress Syndrome of Functional Dyspepsia
Brief Title: International Clinical Study of Zhizhu Kuanzhong Capsule
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017YFC1703703
Record Dates: First submitted 2019-01-28; First posted 2019-01-31 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-01

CONDITIONS: Functional Dyspepsia; Postprandial Distress Syndrome
Keywords: Functional Dyspepsia; Postprandial Distress Syndrome; Traditional Chinese Medicine; efficacy; safety; clinical evaluation

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, multi-center
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zhizhu Kuanzhong Capsule (Experimental): Zhizhu Kuanzhong Capsule Arm is Zhizhu Kuanzhong Capsule, Specification: 0.43 g/granule; Manufacturer: Lonch Group, Shuangren Pharmaceutical Co., Ltd. ; Approval number: NMPA approval number: GUOYAOZHUNZI Z20020003; Dosage and administration: 3 capsules at a time, 3 times a day, taken orally 10-15 min before meals
  Interventions: Drug: Zhizhu Kuanzhong Capsule
- Zhizhu Kuanzhong Placebo Capsule (Placebo Comparator): Zhizhu Kuanzhong Placebo Capsule Arm is Zhizhu Kuanzhong Capsule Mimics composed of microcrystalline cellulose, mannitol and magnesium stearate, which used for filling agent and lubricant respectively; Specification: 0.43 g/granule; Manufacturer: Lonch Group, Shuangren Pharmaceutical Co., Ltd.; Dosage and administration: Be identical with the investigational drug.
  Interventions: Drug: Zhizhu Kuanzhong Placebo Capsule

INTERVENTIONS:
Drug: Zhizhu Kuanzhong Capsule — Zhizhu Kuanzhong Capsule, 3 capsules at a time, 3 times a day, taken orally 10-15 min before meals. an 8-week intervention period
  Other Names: ZZKZ capsule
  Arms: Zhizhu Kuanzhong Capsule
Drug: Zhizhu Kuanzhong Placebo Capsule — Placebo, 3 capsules at a time, 3 times a day, taken orally 10-15 min before meals. an 8-week intervention period
  Other Names: placebo
  Arms: Zhizhu Kuanzhong Placebo Capsule

SUMMARY:
This trial aims to evaluate the clinical efficacy and safety of Zhizhu Kuanzhong Capsule in the treating patients with functional dyspepsia postprandial distress syndrome(FD PDS). Half of participants will receive Zhizhu Kuanzhong Capsule,while the other will receive a placebo.

DETAILED DESCRIPTION:
Functional dyspepsia (FD) is one of the most common functional gastrointestinal disorders. Current data from clinical studies have shown that traditional Chinese medicine can obviously relieve clinical symptoms of patients with FD, and has special advantages and good clinical application prospects in the treatment of FD. Zhizhu Kuanzhong Capsule is mainly composed of the following 4 kinds of Chinese herbs: Rhizoma Atractylodis Macrocephala, Fructus Aurantii Immaturus, Radix Bupleuri and Fructus Crataegi. This trial aims to evaluate the clinical efficacy and safety of Zhizhu Kuanzhong Capsule in the treating patients with functional dyspepsia postprandial distress syndrome(FD PDS). This is a multi-center, stratified-block randomized, double-blind and placebo parallel-controlled trial. The comparison between the investigational drug and the placebo will be conducted with superiority design. About 480 subjects matched Rome IV diagnostic criteria for FD PDS will be enrolled. For each subject, this study includes a 0-2 week screening period, a 1-week run-in period, an 8-week double-blind treatment period, and a 4-week follow-up period. The drugs used in the clinical study (including investigational drug and placebo) will be supplied by Shuangren Pharmaceutical Co., Ltd. of Lonch Group.The quality standards and test methods for the placebo are consistent with those for the investigational drug, and the quality test meets the proposed quality standards. The selection and evaluation bias are controlled by means of strictly implementing randomized control blinded method etc, and the investigator will be trained on the consistency of scale evaluation.The electronic case report form (hereinafter referred to as eCRF) of this trial is created using the Medical Clinical Trial Data Management System (eCDMS3.0) for online data acquisition and management via the Internet. The data in the eCRF are from the original documents such as the original medical records and the physicochemical examination report sheets and should be consistent with the original documents. The response rate for functional dyspepsia VAS score will be compared between the test group and control group at 8 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the Rome IV diagnostic criteria for functional dyspepsia-postprandial distress syndrome;
2. * At least 3 days during the one-week run-in period with VAS score ≥ 4 for major symptoms (at least one of postprandial fullness discomfort and early satiety) .
3. Age between 18 and 65 years old (including 18 and 65 years old), male or female, outpatients;
4. **Be able to discontinue prohibited medications that may affect the evaluation of the effectiveness, such as acid inhibition/antacids, prokinetic agents, non-steroidal anti-inflammatory drugs, anticholinergic agents, glucocorticoids, and therapeutic medication for H. pylori eradication.
5. Each subject is informed and voluntarily signed the informed consent form(ICF).

   * Subjects who entered the one-week run-in period are self-rated on the Visual Analogue Score (VAS) for the degree of discomfort with both symptoms of postprandial fullness and early fullness, with subjects indicating the degree of discomfort on a 10 cm ruler marked 0- "Asymptomatic or No Discomfort"and 10- "Extreme Severe or Extreme Discomfort"at its head and tail, respectively. The rating was made once a day and 7 days a week with scores of 0 to 10.

     * A 2-week wash-out period is required for patients taking prohibited medications prior to screening.

Exclusion Criteria:

1. Gastroscopic findings of gastric cancer, peptic ulcer, erosive gastritis (grade 2 or higher), moderate to severe atrophic gastritis, dysplasia, or other organ gastrointestinal disease.
2. Patients with a history of abdominal surgery (except for appendectomy and cesarean section).
3. Patients with immune system defects (such as leukaemia or cancer), or those who have been administered immunosuppressive agents or glucocorticoids within the past 3 months.
4. Patients who combined severe cardiac and pulmonary insufficiency, insufficiency of liver (ALT/AST > 1.5 times the upper limit of the normal value) and kidney insufficiency (BUN/Serum Creatinine > the upper limit of the normal value), abnormal of endocrine system( such as diabetes and thyroid dysfunction), abnormal hematopoietic system, and iron deficiency anemia as indicated on hematological examination.
5. Patients with severe anxiety and depression.
6. Patients with psychosis and mental retardation as well as language disorder precluding the ability of filling scales or recording symptoms.
7. Pregnant (a female of childbearing potential with a positive pregnancy test) or lactating females; or patients of childbearing potential without effective contraception.
8. Patients who are known to be allergic to the ingredients of this drug.
9. Patients who are suspected to have or indeed have a history of alcohol or drug abuse.
10. Patients who have participated in a clinical trial in the past 3 months.
11. Patients who are deemed by the investigator as being not suitable for participation in the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of the response at 8 weeks after randomization | up to 8 weeks
  Subjects with the functional dyspepsia-postprandial distress syndrome are self-rated on the Visual Analogue Score (VAS) which is a scale of 0-10, with subjects indicating the degree of discomfort on a 10 cm ruler marked 0- "Asymptomatic or No Discomfort "to 10- "Extreme Severe or Extreme Discomfort "at its head and tail, respectively. The record is made once a day and 7 days a week via a diary card. For VAS scores for postprandial fullness discomfort and early satiety, the integral average for both symptoms over the past week is evaluated, and a 50% decrease from baseline in the integral average at 8 Weeks is recorded as a response.

SECONDARY OUTCOMES:
The change of VAS score of each symptom of functional dyspepsia | Up to 8 weeks
  On the diary cards, subjects recorded the Visual Analogue Score (VAS) of each symptom of the functional dyspepsia daily. VAS is scored on a scale of 0-10 which the higher the score, the severer the symptom is. The record is made once a day and 7 days. The investigators use the average of the weekly VAS scores as the symptom intensity score for this week, with one VAS score per week. The change in the score of each symptom at 8 weeks after randomization relative to the baseline is evaluated.
Overall treatment response rate | Up to 8 weeks
  The overall treatment efficacy is evaluated using a 7-point Likert Overall Evaluation Scale (OTE). The clinical investigators asked the subjects the following questions weekly: "In the last week, how much have your dyspeptic symptoms been alleviated as compared to pre-treatment? " There are 7 options: ① the symptoms improved significantly, ② the symptoms improved, ③ the symptoms improved slightly, ④ the symptoms did not change, ⑤ the symptoms aggravated slightly, ⑥ the symptoms aggravated, ⑦ the symptoms aggravated significantly. At the last visit time point of the treatment cycle, patients who selected ① and ② were defined as treatment responders, and those who selected ③-⑦ were defined as non-responders. The response rate at 8 weeks after randomization between the groups are compared for differences.
Short Form Nepean Dyspepsia Index (SFNDI) | Up to 8 weeks
  Short Form-Nepean Dyspepsia Index (SFNDI) is a reliable and valid measure of quality of life in functional dyspepsia with 10 items which questions are about how subjects stomach pain, discomfort, or other epigastric symptoms over the last 14 days affect their lives. Add up the ten items for each of the five sub-scale scores (range of each sub-scale 2-10). The changes of SFNDI score at 4 weeks and 8 weeks after randomization relative to the baseline are calculated.
Hospital Anxiety and Depression Scale score | Up to 8 weeks
  The Hospital Anxiety and Depression Scale (HAD) is mainly used in patients in general hospitals which provides two sets of tests to assess the state of anxiety and depression, respectively. Among them, A stands for anxiety items, D stands for depression items, and each item is scored at four levels. Each of the two sets of items are superimposed to obtain their respective total score. A total score of 0 to 7 indicates normal, 8 to 10 indicates borderline abnormal, and 11 to 21 indicates abnormal. The changes of HAD score at 4 weeks and 8 weeks after randomization relative to the baseline are calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Lu, Md, Phd, Study Director — Xiyuan Hospital of China Academy of Chinese Medical Sciences
Locations (16):
- Princess Alexandra Hospital, Brisbane, Queensland, Australia
- China (15):
  - Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Peking Union Medical College Hospital of Chinese Academy of Medical Sciences, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Hong Kong Baptist University, Hong Kong, Hongokng
  - Wuhan Union Hospital, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - Kulun Qimeng Hospital, Tongliao, Neimenggu
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Affiliated Hospital of Shaanxi University of traditional Chinese medicine, Xi’an, Shanxi
  - Shaanxi Academy of Traditional Chinese Medicine, Xi’an, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiao M, Zhong LLD, Lam WC, Zhao Y, Gwee KA, Holtmann G, Tack J, Suzuki H, Chen MH, Xiao Y, Hou X, Liu J, Li Y, Tang XD, Lu F. Zhizhu Kuanzhong Capsule in treating patients with functional dyspepsia postprandial distress syndrome: study protocol for a multicenter, randomized, double-blind, placebo-controlled, parallel-group clinical trial. Trials. 2022 Jun 2;23(1):454. doi: 10.1186/s13063-022-06396-5. PMID 35655286